CLINICAL TRIAL: NCT00463086
Title: A Randomized-controlled Trial of Isoniazid Plus Highly Active Antiretroviral Therapy Against Placebo to Prevent Tuberculosis in HIV-infected Persons
Brief Title: Isoniazid Plus Antiretroviral Therapy to Prevent Tuberculosis in HIV-infected Persons
Acronym: HAART-IPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other); Imperial College London (Other); Johns Hopkins University (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Prof Gary Maartens, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HAARTIPT07
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Tuberculosis; Latent Tuberculosis Infection; HIV Infections
Keywords: Tuberculosis; TB; Mycobacteria; HIV; Human immunodeficiency virus; Latent tuberculosis infection; HAART; Highly active anti-retroviral therapy; Isoniazid preventive therapy; INH; Opportunistic infections; HIV-1; Treatment Experienced; AIDS; Mycobacterium Tuberculosis
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis; HIV Infections; Mycobacterium Infections; Acquired Immunodeficiency Syndrome; Opportunistic Infections | interventions — Isoniazid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.Isoniazid (INH) (Experimental): A self-administered daily dose of 5mg/kg of Isoniazid (300mg if weight is more than or equal to 50kg and 200mg if weight is less than 50kg)
  Interventions: Drug: isoniazid
- 2. Placebo (Placebo Comparator): A self-administered daily dose of 5mg/kg of placebo for 12months (300mg if weight is more than or equal to 50kg and 200mg if weight is less than 50kg)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: isoniazid — A self-administered daily dose of 5mg/kg of Isoniazid or placebo for 12months(300mg if weight is more than or equal to 50kg and 200mg if weight is less than 50kg)
  Arms: 1.Isoniazid (INH)
Drug: Placebo — A self-administered dose of 5mg/kg of placebo (300mg if weight is more than or equal to 50kg and 200mg if weight is less than 50kg)
  Arms: 2. Placebo

SUMMARY:
The purpose of this study is to evaluate whether isoniazid can safely (and further) reduce the risk of tuberculosis in HIV infected people receiving HAART.

DETAILED DESCRIPTION:
The incidence of Tuberculosis (TB) in poor settlements around Cape Town continues to rise despite highly-active-anti-retroviral therapy (HAART) roll-out and DOTS. In Khayelitsha district, where this project will be conducted, TB incidence is about 1600/100000. There is an equally high HIV prevalence, currently 33%. Over 50% of adults presenting with active TB are co-infected with HIV and a third of all patients starting HAART have active TB. Although HAART has been shown to reduce the overall risk of TB by 59-80%, this risk still far exceeds the general risk. In the Khayelitsha HAART cohort, the risk of developing TB whilst on HAART is ~12 per 100 p-y. In the nearby community of Gugulethu, there is a 14% risk of active TB with at least half of the cases occurring within the first 3months on HAART. In a region where RD1-detected prevalence of latent TB infection is at least 80%, there is a real concern that TB will likely undo the benefit of HAART in the long run. Additional measures are therefore required to reduce the risk of TB in those already receiving or starting HAART. Isoniazid preventive therapy (IPT) represents an option but there is insufficient evidence to determine whether IPT can further (and safely) reduce the risk of TB in the HAART era. In a RCT, we propose to evaluate whether IPT can reduce the risk of active TB in patients receiving HAART.

A total minimum sample size of 1204 is required for the study to detect a 35% reduction in the hazard rates for tuberculosis in the intervention group (h1= 0.052) compared to the control group (h0=0.085) at a power of 80% and a Type II error of 0.05. Our maximum targeted sample size when losses to follow-up and subgroup analyses are considered is 1445. Development of TB will be the primary endpoint.

Additional information (on 10 August 2010):

Recruitment and enrolment into the study was completed in October 2009. We have screened over 2000 patients already on ART and those newly starting ART. However, instead of enrolling our desired maximum sample size of 1445, a revised minimum total of 1368 were instead randomized to the study drug. This followed an amendment to the sample size necessitated by new information on the clinical site; primarily higher rates of patients lost to follow-up at the clinical site than previously anticipated. The amendment to our sample size was reported to, and acknowledged by, the Research Ethics Committee of the University of Cape Town. Follow-up of participants will continue until Oct/November 2011.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female attendees (age ≥18yo) of the Ubuntu HIV and ARV Clinic identified as eligible for the ARV programme will be invited to participate.
2. Willingness to participate
3. Able to engage in informed consent procedures

Exclusion Criteria:

1. Evidence of active TB or suspicion of active TB as determined by a symptoms screening algorithm.
2. Current TB chemotherapy ( TB treatment completed in the preceding 30 days will not be an exclusion)
3. Current or previous treatment of latent TB infection since HIV infection (any duration)
4. Current treatment with fluoroquinolones or other antibiotics with significant anti-tuberculous activity currently being used to treat TB in South Africa
5. Past reaction/intolerance to INH.
6. Acute hepatitis or existing Grade III-IV peripheral neuropathy.
7. Pregnancy or < 6weeks post-partum period (Due to increased risk of hepatotoxicity).
8. Grade III or higher baseline abnormal liver function. (Note: toxicity grades are all according to ACTG toxicity tables for persons on ART).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1368 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Rate of development of TB (microbiologically confirmed TB or highly probable TB) during the 36 month risk period | Patients are assessed for TB one two monthly at each ART re-fill appointment

SECONDARY OUTCOMES:
Rate of drug toxicity (specifically, peripheral neuropathy, hepatitis +/-raised ALT grade III or worse and allergic rashes grade III or worse | during the intervention period (ALT determined at baseline, 1, 2 and 3 months and then 3-monthly. the last safety determination is at 12 months post initiation of the study drug)
Proportions adhering to study drug and HAART at the end of each study year as measured by pharmacy refills | 1 month to two monthly, depending on the individual patient's clinic appointment
Rate of development of INH monoresistance during the 36 month risk period. | 36 months
Death | 36 months
Worsening ART outcomes (virological and immunological failure) | CD4+count and viral load are assessed as per clinic protocol (6 monthly post ART initiation)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Maartens (overall PI), FCP, Principal Investigator — University of Cape Town; Eric Goemaere (co-investigator), MBBS, Study Director — Medecins Sans Frontieres, Netherlands; Molebogeng X Rangaka (Lead Investigator), MBChB, Study Director — University of Cape Town; Gilles van Cutsem co-investigator), MBBS, Study Director — Medecins Sans Frontieres, Netherlands; Andrew Boulle co-investigator), FCP, Study Director — University of Cape Town; Robert J Wilkinson (PI:Immunology Studies), FRCP, Study Director — Wellcome Trust; Shahied Mathee (Ubuntu PMO), MBChB, Study Director — Provincial Government of Western Cape
Locations (1):
- Ubuntu Clinic,Site B Khayelitsha, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Rangaka MX, Wilkinson RJ, Boulle A, Glynn JR, Fielding K, van Cutsem G, Wilkinson KA, Goliath R, Mathee S, Goemaere E, Maartens G. Isoniazid plus antiretroviral therapy to prevent tuberculosis: a randomised double-blind, placebo-controlled trial. Lancet. 2014 Aug 23;384(9944):682-90. doi: 10.1016/S0140-6736(14)60162-8. Epub 2014 May 13. PMID 24835842